CLINICAL TRIAL: NCT01055093
Title: Prospective Study on Diabetes Mellitus and Its Complications in Newly Diagnosed Adult Patients
Acronym: GDC
Status: Recruiting | Type: Observational
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: GDC-Study-01
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: diabetes mellitus; prospective observational study; diabetic complications
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, PBMC, serum, plasma, urine, stool
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Diabetes Cohort: Prospectively followed cohort of newly diagnosed patients with diabetes mellitus, aged 18-69 years at inclusion into the study
- Control Cohort: Prospectively followed cohort of glucose tolerant humans, aged 18-69 years at inclusion into the study

SUMMARY:
The aim of the prospective observational GDC-Study in patients with newly diagnosed diabetes mellitus aged 18-69 years at inclusion into the study is to characterize in detail the clinical, metabolical and immunological phenotype and monitor the progression of the disease and to compare the phenotype to glucose tolerant humans of similar age, body mass and sex distribution.

DETAILED DESCRIPTION:
In detail, the following questions will be answered:

1. Are there different phenotypes with respect to insulin secretion, insulin sensitivity, micro- and macrovascular status and diabetic neuropathy at time of diagnosis?
2. Which factors modify the progression of the disease (Nutrition, subclinical inflammation, energy metabolism and physical activity)?
3. Can we identify subgroups at baseline with different progression of the disease? Patients are thoroughly examined at baseline and after 2, 5, and 10 years with annual telephone contacts in between.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes mellitus according to ADA criteria
* Age 18-69
* Diabetes duration since diagnosis < 12 months
* Control cohort: proven normal glucose tolerance according to ADA criteria

Exclusion Criteria:

* Diabetes mellitus category 3 B-H (ADA criteria)
* Pregnancy
* Severe renal, liver or heart disease
* malignant cancer
* severe psychiatric illness or addiction
* participation in an intervention trial

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from the general populations by screening
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2005-09 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2040-09 (Estimated)

PRIMARY OUTCOMES:
Change of insulin sensitivity (M-Value) | 2 and 5 years
  measurement of whole body insulin sensitivity with hyperinsulinamic euglicamic clamp

SECONDARY OUTCOMES:
Change of insulin secretion | 2 and 5 years
  measurement of insulin secretion with glucagon test, mixed-meal test and intravenous glucose tolerance test
Incidence of any diabetic complication | 2-10 years
  The prevalence of diabetic complications

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Szendroedi J, Saxena A, Weber KS, Strassburger K, Herder C, Burkart V, Nowotny B, Icks A, Kuss O, Ziegler D, Al-Hasani H, Mussig K, Roden M; GDS Group. Cohort profile: the German Diabetes Study (GDS). Cardiovasc Diabetol. 2016 Apr 7;15:59. doi: 10.1186/s12933-016-0374-9. PMID 27053136
- [Background] Kossler T, Bobrov P, Strassburger K, Kuss O, Zaharia OP, Karusheva Y, Moser C, Bodis K, Burkart V, Roden M, Szendroedi J; GDS Group. Impact of mixed meal tolerance test composition on measures of beta-cell function in type 2 diabetes. Nutr Metab (Lond). 2021 May 4;18(1):47. doi: 10.1186/s12986-021-00556-1. PMID 33947421
- [Background] Kupriyanova Y, Zaharia OP, Bobrov P, Karusheva Y, Burkart V, Szendroedi J, Hwang JH, Roden M; GDS group. Early changes in hepatic energy metabolism and lipid content in recent-onset type 1 and 2 diabetes mellitus. J Hepatol. 2021 May;74(5):1028-1037. doi: 10.1016/j.jhep.2020.11.030. Epub 2020 Nov 28. PMID 33259845
- [Background] Zaharia OP, Strassburger K, Knebel B, Kupriyanova Y, Karusheva Y, Wolkersdorfer M, Bodis K, Markgraf DF, Burkart V, Hwang JH, Kotzka J, Al-Hasani H, Szendroedi J, Roden M; GDS Group. Role of Patatin-Like Phospholipase Domain-Containing 3 Gene for Hepatic Lipid Content and Insulin Resistance in Diabetes. Diabetes Care. 2020 Sep;43(9):2161-2168. doi: 10.2337/dc20-0329. Epub 2020 Jun 19. PMID 32910776
- [Background] Maalmi H, Herder C, Strassburger K, Urner S, Jandeleit-Dahm K, Zaharia OP, Karusheva Y, Bongaerts BWC, Rathmann W, Burkart V, Szendroedi J, Roden M. Biomarkers of Inflammation and Glomerular Filtration Rate in Individuals with Recent-Onset Type 1 and Type 2 Diabetes. J Clin Endocrinol Metab. 2020 Dec 1;105(12):dgaa622. doi: 10.1210/clinem/dgaa622. PMID 32879938
- [Background] Kanti G, Anadol-Schmitz E, Bobrov P, Strassburger K, Kahl S, Zaharia OP, Sarabhai T, Karusheva Y, Burkart V, Markgraf DF, Trenkamp S, Ziegler D, Szendroedi J, Roden M; GDS Group. Vitamin B12 and Folate Concentrations in Recent-onset Type 2 Diabetes and the Effect of Metformin Treatment. J Clin Endocrinol Metab. 2020 Jun 1;105(6):dgaa150. doi: 10.1210/clinem/dgaa150. PMID 32219330
- [Background] Bodis K, Jelenik T, Lundbom J, Markgraf DF, Strom A, Zaharia OP, Karusheva Y, Burkart V, Mussig K, Kupriyanova Y, Ouni M, Wolkersdorfer M, Hwang JH, Ziegler D, Schurmann A, Roden M, Szendroedi J; GDS Study Group. Expansion and Impaired Mitochondrial Efficiency of Deep Subcutaneous Adipose Tissue in Recent-Onset Type 2 Diabetes. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1331-43. doi: 10.1210/clinem/dgz267. PMID 31838512
- [Background] Puttgen S, Bonhof GJ, Strom A, Mussig K, Szendroedi J, Roden M, Ziegler D. Augmented Corneal Nerve Fiber Branching in Painful Compared With Painless Diabetic Neuropathy. J Clin Endocrinol Metab. 2019 Dec 1;104(12):6220-6228. doi: 10.1210/jc.2019-01072. PMID 31390004
- [Background] Zaharia OP, Strassburger K, Strom A, Bonhof GJ, Karusheva Y, Antoniou S, Bodis K, Markgraf DF, Burkart V, Mussig K, Hwang JH, Asplund O, Groop L, Ahlqvist E, Seissler J, Nawroth P, Kopf S, Schmid SM, Stumvoll M, Pfeiffer AFH, Kabisch S, Tselmin S, Haring HU, Ziegler D, Kuss O, Szendroedi J, Roden M; German Diabetes Study Group. Risk of diabetes-associated diseases in subgroups of patients with recent-onset diabetes: a 5-year follow-up study. Lancet Diabetes Endocrinol. 2019 Sep;7(9):684-694. doi: 10.1016/S2213-8587(19)30187-1. Epub 2019 Jul 22. PMID 31345776
- [Background] Simon MC, Moller-Horigome A, Strassburger K, Nowotny B, Knebel B, Mussig K, Herder C, Szendroedi J, Roden MW; German Diabetes Study Group. Correlates of Insulin-Stimulated Glucose Disposal in Recent-Onset Type 1 and Type 2 Diabetes. J Clin Endocrinol Metab. 2019 Jun 1;104(6):2295-2304. doi: 10.1210/jc.2018-02057. PMID 30689904
- [Background] Rathmann W, Strassburger K, Bongaerts B, Kuss O, Mussig K, Burkart V, Szendroedi J, Kotzka J, Knebel B, Al-Hasani H, Roden M; GDS Group. A variant of the glucose transporter gene SLC2A2 modifies the glycaemic response to metformin therapy in recently diagnosed type 2 diabetes. Diabetologia. 2019 Feb;62(2):286-291. doi: 10.1007/s00125-018-4759-z. Epub 2018 Nov 9. PMID 30413829
- [Background] Grobosch S, Kuske S, Linnenkamp U, Ernstmann N, Stephan A, Genz J, Begun A, Haastert B, Szendroedi J, Mussig K, Burkart V, Roden M, Icks A; GDS Group. What information needs do people with recently diagnosed diabetes mellitus have and what are the associated factors? A cross-sectional study in Germany. BMJ Open. 2018 Oct 31;8(10):e017895. doi: 10.1136/bmjopen-2017-017895. PMID 30385437
- [Background] Schroder K, Szendroedi J, Benthin A, Gontscharuk V, Ackermann P, Volker M, Steingrube N, Nowotny B, Ziegler D, Mussig K, Geerling G, Kuss O, Roden M, Guthoff R; GDS Cohort. German Diabetes Study - Baseline data of retinal layer thickness measured by SD-OCT in early diabetes mellitus. Acta Ophthalmol. 2019 Mar;97(2):e303-e307. doi: 10.1111/aos.13851. Epub 2018 Sep 21. PMID 30238609
- [Background] van Gemert T, Wolwer W, Weber KS, Hoyer A, Strassburger K, Bohnau NT, Bruggen MA, Ovelgonne K, Gossmann EM, Burkart V, Szendroedi J, Roden M, Mussig K; GDS Group. Cognitive Function Is Impaired in Patients with Recently Diagnosed Type 2 Diabetes, but Not Type 1 Diabetes. J Diabetes Res. 2018 Aug 9;2018:1470476. doi: 10.1155/2018/1470476. eCollection 2018. PMID 30159333
- [Background] Ziegler D, Strom A, Kupriyanova Y, Bierwagen A, Bonhof GJ, Bodis K, Mussig K, Szendroedi J, Bobrov P, Markgraf DF, Hwang JH, Roden M; GDS Group. Association of Lower Cardiovagal Tone and Baroreflex Sensitivity With Higher Liver Fat Content Early in Type 2 Diabetes. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1130-1138. doi: 10.1210/jc.2017-02294. PMID 29267946
- [Background] Zaharia OP, Bobrov P, Strassburger K, Bodis K, Karusheva Y, Scholz M, Markgraf DF, Burkart V, Schloot NC, Mussig K, Szendroedi J, Roden M; GDS Group. Metabolic Characteristics of Recently Diagnosed Adult-Onset Autoimmune Diabetes Mellitus. J Clin Endocrinol Metab. 2018 Feb 1;103(2):429-437. doi: 10.1210/jc.2017-01706. PMID 29220505
- [Background] Rohling M, Strom A, Bonhof G, Puttgen S, Bodis K, Mussig K, Szendrodi J, Markgraf D, Lehr S, Roden M, Ziegler D; German Diabetes Study Group. Differential Patterns of Impaired Cardiorespiratory Fitness and Cardiac Autonomic Dysfunction in Recently Diagnosed Type 1 and Type 2 Diabetes. Diabetes Care. 2017 Feb;40(2):246-252. doi: 10.2337/dc16-1898. Epub 2016 Nov 29. PMID 27899499
- [Background] Weber KS, Strassburger K, Pacini G, Nowotny B, Mussig K, Szendroedi J, Herder C, Roden M; German Diabetes Study group. Circulating adiponectin concentration is inversely associated with glucose tolerance and insulin secretion in people with newly diagnosed diabetes. Diabet Med. 2017 Feb;34(2):239-244. doi: 10.1111/dme.13278. Epub 2016 Nov 17. PMID 27770592
- [Background] Weber KS, Knebel B, Strassburger K, Kotzka J, Stehle P, Szendroedi J, Mussig K, Buyken AE, Roden M; GDS Group. Associations between explorative dietary patterns and serum lipid levels and their interactions with ApoA5 and ApoE haplotype in patients with recently diagnosed type 2 diabetes. Cardiovasc Diabetol. 2016 Sep 27;15(1):138. doi: 10.1186/s12933-016-0455-9. PMID 27677442
- [Background] Apostolopoulou M, Strassburger K, Herder C, Knebel B, Kotzka J, Szendroedi J, Roden M; GDS group. Metabolic flexibility and oxidative capacity independently associate with insulin sensitivity in individuals with newly diagnosed type 2 diabetes. Diabetologia. 2016 Oct;59(10):2203-7. doi: 10.1007/s00125-016-4038-9. Epub 2016 Jul 4. PMID 27376543
- [Background] Gancheva S, Bierwagen A, Kaul K, Herder C, Nowotny P, Kahl S, Giani G, Klueppelholz B, Knebel B, Begovatz P, Strassburger K, Al-Hasani H, Lundbom J, Szendroedi J, Roden M; German Diabetes Study (GDS) Group. Variants in Genes Controlling Oxidative Metabolism Contribute to Lower Hepatic ATP Independent of Liver Fat Content in Type 1 Diabetes. Diabetes. 2016 Jul;65(7):1849-57. doi: 10.2337/db16-0162. Epub 2016 Apr 19. PMID 27207512
- [Background] Knebel B, Strassburger K, Szendroedi J, Kotzka J, Scheer M, Nowotny B, Mussig K, Lehr S, Pacini G, Finner H, Kluppelholz B, Giani G, Al-Hasani H, Roden M; German Diabetes Study Group. Specific Metabolic Profiles and Their Relationship to Insulin Resistance in Recent-Onset Type 1 and Type 2 Diabetes. J Clin Endocrinol Metab. 2016 May;101(5):2130-40. doi: 10.1210/jc.2015-4133. Epub 2016 Feb 1. PMID 26829444
- [Background] Weber KS, Nowotny B, Strassburger K, Pacini G, Mussig K, Szendroedi J, Herder C, Roden M; GDS Group. The Role of Markers of Low-Grade Inflammation for the Early Time Course of Glycemic Control, Glucose Disappearance Rate, and beta-Cell Function in Recently Diagnosed Type 1 and Type 2 Diabetes. Diabetes Care. 2015 Sep;38(9):1758-67. doi: 10.2337/dc15-0169. Epub 2015 Jul 7. PMID 26153272
- [Background] Menart-Houtermans B, Rutter R, Nowotny B, Rosenbauer J, Koliaki C, Kahl S, Simon MC, Szendroedi J, Schloot NC, Roden M; German Diabetes Study Group. Leukocyte profiles differ between type 1 and type 2 diabetes and are associated with metabolic phenotypes: results from the German Diabetes Study (GDS). Diabetes Care. 2014 Aug;37(8):2326-33. doi: 10.2337/dc14-0316. PMID 25061140
- [Derived] Trinks N, Putzer J, Sutkowski A, Burkart V, Roden M, Kuss O. Comparison of Vyntus CPX and Vmax Encore 29N for indirect calorimetry: a randomised crossover study in participants of the German Diabetes Study with type 2 diabetes. BMJ Open. 2025 Dec 10;15(12):e104761. doi: 10.1136/bmjopen-2025-104761. PMID 41371739
- [Derived] Jonuscheit M, Korzekwa B, Schar M, Mevenkamp J, Wierichs S, Bobrov P, Sarabhai T, Kahl S, Roden M, Schrauwen-Hinderling VB. 31P-MRS saturation transfer for assessing human hepatic ATP synthesis at clinical field strength. Eur Radiol Exp. 2025 May 13;9(1):51. doi: 10.1186/s41747-025-00588-9. PMID 40360906
- [Derived] Kaya S, Khamees A, Geerling G, Strzalkowski P, Gontscharuk V, Szendroedi J, Mussig K, Ziegler D, Roden M, Guthoff R; GDS Cohort. Macular perfusion alterations in people with recent-onset diabetes and novel diabetes subtypes. Diabetologia. 2025 Jun;68(6):1140-1156. doi: 10.1007/s00125-025-06407-5. Epub 2025 Mar 31. PMID 40164944
- [Derived] Kupriyanova Y, Yurchenko I, Bobrov P, Bartels F, Wierichs S, Jonuscheit M, Korzekwa B, Prystupa K, Schon M, Mendez D, Trenkamp S, Burkart V, Wagner R, Schrauwen-Hinderling V, Roden M; German Diabetes Study (GDS) Group. Alterations of hepatic lipid content following COVID-19 in persons with type 2 diabetes. BMJ Open Diabetes Res Care. 2025 Feb 18;13(1):e004727. doi: 10.1136/bmjdrc-2024-004727. PMID 39965871
- [Derived] Spagnuolo MC, Gottmann P, Sommer J, Borgmann SO, Strassburger K, Rathmann W, Zaharia OP, Trenkamp S, Wagner R, Icks A, Herder C, Roden M, Maalmi H; GDS Group. Three-protein signature is associated with baseline and persistently elevated or recurrent depressive symptoms in individuals with recent-onset diabetes. BMJ Open Diabetes Res Care. 2025 Feb 18;13(1):e004396. doi: 10.1136/bmjdrc-2024-004396. PMID 39965868
- [Derived] Weber KS, Schlesinger S, Goletzke J, Strassburger K, Zaharia OP, Trenkamp S, Wagner R, Lieb W, Buyken AE, Roden M, Herder C; GDS group. Associations of carbohydrate quality and cardiovascular risk factors vary among diabetes subtypes. Cardiovasc Diabetol. 2025 Feb 6;24(1):53. doi: 10.1186/s12933-025-02580-4. PMID 39915806
- [Derived] Weber KS, Schlesinger S, Lang A, Strassburger K, Maalmi H, Zhu A, Zaharia OP, Strom A, Bonhof GJ, Goletzke J, Trenkamp S, Wagner R, Buyken AE, Lieb W, Roden M, Herder C; GDS group. Association of dietary patterns with diabetes-related comorbidities varies among diabetes endotypes. Nutr Metab Cardiovasc Dis. 2024 Apr;34(4):911-924. doi: 10.1016/j.numecd.2023.12.026. Epub 2024 Jan 5. PMID 38418350
- [Derived] Heilmann G, Trenkamp S, Moser C, Bombrich M, Schon M, Yurchenko I, Strassburger K, Rodriguez MM, Zaharia OP, Burkart V, Wagner R, Roden M. Precise glucose measurement in sodium fluoride-citrate plasma affects estimates of prevalence in diabetes and prediabetes. Clin Chem Lab Med. 2023 Oct 24;62(4):762-769. doi: 10.1515/cclm-2023-0770. Print 2024 Mar 25. PMID 37870928
- [Derived] Baechle C, Lang A, Strassburger K, Kuss O, Burkart V, Szendroedi J, Mussig K, Weber KS, Schrauwen-Hinderling V, Herder C, Roden M, Schlesinger S; GDS group. Association of a lifestyle score with cardiometabolic markers among individuals with diabetes: a cross-sectional study. BMJ Open Diabetes Res Care. 2023 Jul;11(4):e003469. doi: 10.1136/bmjdrc-2023-003469. PMID 37433698
- [Derived] Goletzke J, Weber KS, Kossler T, Zaharia OP, Bodis K, Mussig K, Szendroedi J, Burkart V, Stutz B, Nothlings U, Buyken AE, Roden M; GDS Group. Relative validity of a glycemic index extended food-frequency questionnaire. Nutr Metab Cardiovasc Dis. 2022 Oct;32(10):2310-2320. doi: 10.1016/j.numecd.2022.07.007. Epub 2022 Jul 16. PMID 35973887
- [Derived] Zaharia OP, Schon M, Loffler L, Strassburger K, Moser C, Yurchenko I, Bodis K, Antoniou S, Karusheva Y, Szendroedi J, Burkart V, Roden M. Metabolic Factors Predict Changes in Endothelial Function During the Early Course of Type 1 and Type 2 Diabetes. J Clin Endocrinol Metab. 2022 Sep 28;107(10):e4167-e4176. doi: 10.1210/clinem/dgac480. PMID 35965389
- [Derived] Bodis K, Knebel B, Nowotny B, Bobrov P, Kupriyanova Y, Zaharia OP, Karusheva Y, Schon M, Wolkersdorfer M, Burkart V, Al-Hasani H, Markgraf D, Mussig K, Roden M, Szendroedi J; GDS study group. Hepatic energy metabolism in a family with a glucokinase gene mutation and dysglycemia. Diabetes Res Clin Pract. 2022 Mar;185:109779. doi: 10.1016/j.diabres.2022.109779. Epub 2022 Feb 14. PMID 35176401
- [Derived] Saatmann N, Zaharia OP, Strassburger K, Pesta DH, Burkart V, Szendroedi J, Gerdes N, Kelm M, Roden M. Physical Fitness and Cardiovascular Risk Factors in Novel Diabetes Subgroups. J Clin Endocrinol Metab. 2022 Mar 24;107(4):1127-1139. doi: 10.1210/clinem/dgab810. PMID 34748634
- [Derived] Pesta D, Jelenik T, Zaharia OP, Bobrov P, Gorgens S, Bodis K, Karusheva Y, Krako Jakovljevic N, Lalic NM, Markgraf DF, Burkart V, Mussig K, Knebel B, Kotzka J, Eckel J, Strassburger K, Szendroedi J, Roden M. NDUFB6 Polymorphism Is Associated With Physical Activity-Mediated Metabolic Changes in Type 2 Diabetes. Front Endocrinol (Lausanne). 2021 Sep 24;12:693683. doi: 10.3389/fendo.2021.693683. eCollection 2021. PMID 34659107
- [Derived] Zaharia OP, Pesta DH, Bobrov P, Kupriyanova Y, Herder C, Karusheva Y, Bodis K, Bonhof GJ, Knitza J, Simon D, Kleyer A, Hwang JH, Mussig K, Ziegler D, Burkart V, Schett G, Roden M, Szendroedi J. Reduced Muscle Strength Is Associated With Insulin Resistance in Type 2 Diabetes Patients With Osteoarthritis. J Clin Endocrinol Metab. 2021 Mar 25;106(4):1062-1073. doi: 10.1210/clinem/dgaa912. PMID 33382877
- [Derived] Eckstein ML, Farinha JB, McCarthy O, West DJ, Yardley JE, Bally L, Zueger T, Stettler C, Boff W, Reischak-Oliveira A, Riddell MC, Zaharieva DP, Pieber TR, Muller A, Birnbaumer P, Aziz F, Brugnara L, Haahr H, Zijlstra E, Heise T, Sourij H, Roden M, Hofmann P, Bracken RM, Pesta D, Moser O. Differences in Physiological Responses to Cardiopulmonary Exercise Testing in Adults With and Without Type 1 Diabetes: A Pooled Analysis. Diabetes Care. 2021 Jan;44(1):240-247. doi: 10.2337/dc20-1496. Epub 2020 Nov 12. PMID 33184152
- See also: Official website of the German Diabetes Center — https://ddz.de/